CLINICAL TRIAL: NCT06969495
Title: A Clinical Investigation Into the Dermal Application of L. Rhinocerus TM02(r) Water Extract for Mouth Ulceration
Brief Title: Pilot Clinical Study Testing Tiger Milk Mushroom Gel (Lignosus Rhinocerus TM02®) for Treating Mouth Ulcers
Acronym: DERMAL-LR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahsa University (Other)
Responsible Party: Principal Investigator, Yeannie Yap, Senior Lecturer, Mahsa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RP185_05/22
Record Dates: First submitted 2025-04-28; First posted 2025-05-14 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Mouth Ulcer
Keywords: Tiger Milk Mushroom; Mouth ulcers; Wound healing; Natural remedies
MeSH Terms: conditions — Oral Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Base formulation (Placebo Comparator): Participants will receive an oral gel base formulation without the Lignosus rhinocerus extract. The placebo gel will be applied to the mouth ulcer three times daily for seven days.
  Interventions: Other: Placebo
- xLr oral gel (Experimental): Participants will receive an oral gel containing 25% Lignosus rhinocerus TM02® cold water extract (xLr®). The gel will be applied to the mouth ulcer three times daily for seven days.
  Interventions: Other: xLr oral gel
- Kanolone Oral Base Paste (Active Comparator): Participants will receive Kanolone Oral Base Paste (Triamcinolone acetonide 0.1%), a standard topical corticosteroid treatment for aphthous ulcers. The paste will be applied to the mouth ulcer three times daily for seven days.
  Interventions: Drug: Kanolone

INTERVENTIONS:
Other: xLr oral gel — 25% of Cold water extract of Tiger milk mushroom sclerotial powder in a gel form containing xanthan gum as a thickening agent and 0.5% sodium benzoate as a preservative.
  Other Names: TM02 gel
  Arms: xLr oral gel
Other: Placebo — oral gel base formulation without the Lignosus rhinocerus extract
  Other Names: Vehicle ctrl
  Arms: Base formulation
Drug: Kanolone — Kanolone Oral Base Paste (Triamcinolone acetonide 0.1%)
  Other Names: Positive ctrl
  Arms: Kanolone Oral Base Paste

SUMMARY:
This is a pilot clinical trial study to investigate the wound healing capability of a TM02® water extract formulation in patient with minor oral ulcers (2 - 5 mm in size). The sclerotium of L. rhinocerus is traditionally used as a health tonic or treatment regime for asthma, bronchitis, various cancer ailments as well as discomforts caused by fright, fever, cough, vomiting, and injury. Further on to that, this mushroom has also been traditionally used by the local Malay and Chinese communities to treat wounds, although it is yet to be scientifically validated. Its sclerotia are being consumed in the form of decoction, in a betel quid, and other preparation method where the sclerotium is pounded with raw rice, infused, and subsequently taken as a drink. There is also a practice of biting/chewing of the sclerotium by local indigenous communities during their journeys in the wild.

DETAILED DESCRIPTION:
Project overview Lignosus rhinocerus, commonly known as tiger milk mushroom (TMM), is a medicinal fungus native to Southeast Asia. Traditionally, it has been utilized for various health conditions, including wound healing. Recent studies have highlighted its anti-inflammatory, antimicrobial, and immunomodulatory properties, particularly in its cultivated form, TM02® .

Aphthous ulcers, or recurrent aphthous stomatitis (RAS), are common, painful lesions of the oral mucosa affecting a significant portion of the adult population. Current treatments primarily involve topical corticosteroids, which may have side effects with prolonged use. Given the traditional use of L. rhinocerus in wound care, this study aims to evaluate the efficacy of TM02® gel in treating minor oral aphthous ulcers.

Hypothesis and general objective Hypothesis: L. rhinocerus cultivar TM02® gel accelerates the healing process of minor oral aphthous ulcers compared to standard treatments.

Primary Objective: To assess the efficacy of L. rhinocerus TM02® gel in promoting the healing of minor oral aphthous ulcers.

Methodology Mushroom Material and Gel Formulation Lignosus rhinocerus TM02® freeze-dried sclerotia powder (TM02®) was obtained from LiGNO Biotech Sdn. Bhd. (Selangor, Malaysia). This commercially available product is officially registered under the Protection of New Plant Varieties Act (NPVA), Malaysia (Registration No.: PVBT010/11). The authenticity of TM02® was confirmed via polymerase chain reaction (PCR) amplification and sequencing of the internal transcribed spacer (ITS) region. To extract its bioactive compounds, the sclerotia powder underwent cold water extraction at a 1:20 ratio of powder to distilled water, followed by centrifugation and freeze-drying. The resulting extract, referred to as xLr®, was then formulated into an oral gel by incorporating it with xanthan gum as a thickening agent and 0.5% sodium benzoate as a preservative. The final gel formulation (containing 25% xLr®) was stored at room temperature until further use.

Study Design and Ethical Approval A double-blinded, randomised clinical trial was conducted with approval from the Research Management Centre, MAHSA University (Ethics No.: RMC/EC45/2022). Prior to enrolment, all participants received a patient information sheet detailing the study objectives, procedures, potential risks, and benefits. Informed consent was obtained from each participant before proceeding. Systemically healthy patients presenting with minor, isolated aphthous ulcers were recruited, while individuals taking medication, using mouthwash, or consuming herbal products were excluded. A third party managed the randomisation process to ensure impartiality, and both investigators and participants remained blinded to the assigned treatments. For participants with language barriers, a student translator assisted in explaining the study details and consent process to ensure clear communication. All study procedures were conducted in accordance with ethical guidelines and clinical protocols.

Treatment Protocol A total of 21 patients (8 males, 13 females), aged 20-50 years, were randomly allocated into three groups. The control group received the base formulation without xLr®, the test group received the xLr® oral gel, and the standard treatment group was given Kanolone Oral Base Paste (Triamcinolone acetonide 0.1%). Patients were instructed to apply a thin layer of the assigned gel to the ulcer using a dry cotton bud three times daily for seven days, ensuring no eating or drinking for at least 30 minutes post-application.

Clinical Evaluations Pain levels were recorded daily for seven days using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst pain). Ulcer size was measured on Days 1, 3, 5, and 7 using a transparent grid overlay. Each square on the grid represented a surface area of 4 mm². The total ulcer area (mm²) was determined by counting the number of squares within the ulcer's outline, providing an objective assessment of wound size over time. Wound epithelialisation was assessed on Days 3, 5, and 7 by applying a 3% hydrogen peroxide (H₂O₂) solution to the ulcer site. Bubble formation indicated incomplete epithelialisation, whereas the absence of bubbles signified complete epithelialisation, providing a clear and reliable measure of the healing process over time. For cases where epithelialisation required more than seven days-exceeding the study's observation period-it was assigned a value of 8 for analytical consistency.

Study Site The trial was conducted at MAHSA University's clinical facilities, specifically within the Faculty of Dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged between 20 and 50 years
* No history of systemic diseases such as leukemia, hemophilia, uncontrolled diabetes mellitus, or serious cardiac conditions
* Presence of minor oral aphthous ulcers ranging from 2 to 5 mm in size
* No use of medications, including topical steroids or mouthwashes, for at least 3 months prior to the study
* Willingness to provide written informed consent and adhere to the study protocol.

Exclusion Criteria:

* Pregnant or lactating women; Known allergies to any components of the study formulations
* Any condition that, in the opinion of the investigator, may interfere with the study objectives or participant safety.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Pain Assessment | Daily assessments on Days 1 through 7 during the intervention
  Pain levels were assessed daily over a seven-day period using the Visual Analog Scale (VAS), where 0 represented no pain and 10 indicated the worst possible pain.
Wound Epithelialization | Assessments on Days 3, 5, and 7 during the intervention
  Wound epithelialisation was evaluated on Days 3, 5, and 7 by applying a 3% hydrogen peroxide (H₂O₂) solution to the ulcer site. The formation of bubbles indicated incomplete epithelialisation, while the absence of bubbles signified complete epithelialisation, offering a reliable and consistent measure of the healing process.
Ulcer size | Days 1, 3, 5, and 7 during the intervention
  Ulcer size was measured on Days 1, 3, 5, and 7 using a transparent grid overlay. Each square on the grid represented a surface area of 4 mm². The total ulcer area (mm²) was determined by counting the number of squares within the ulcer's outline, providing an objective assessment of wound size over time

CONTACTS AND LOCATIONS:
Locations (1):
- MAHSA University Dental Clinic, Jenjarum, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No